CLINICAL TRIAL: NCT04811625
Title: A Randomized, Open-label, 2-way Crossover Pharmacodynamic and Pharmacokinetic Study of a Novel Pharmaceutical Lipid-aspirin Complex Formulation (PL-ASA) at an 81 mg Dose
Brief Title: Pharmacodynamic and Pharmacokinetic Study of PL-ASA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PL-ASA-010
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PL-ASA capsule, then EC-ASA tablet (Other): PL-ASA capsule 81 mg, then crossover to EC-ASA tablet 81 mg
  Interventions: Drug: PL-ASA
- EC-ASA tablet, then PL-ASA capsule (Active Comparator): EC-ASA tablet 81 mg, then crossover to PL-ASA capsule 81 mg
  Interventions: Drug: PL-ASA

INTERVENTIONS:
Drug: PL-ASA — Pharmacologic profile of different aspirin formulations
  Other Names: Enteric-coated Aspirin (EC-ASA)

SUMMARY:
A randomized, open-label, 2-way crossover pharmacodynamic and pharmacokinetic study of a novel pharmaceutical lipid-aspirin complex formulation (PL-ASA) at an 81 mg dose

DETAILED DESCRIPTION:
This study is a randomized, open-label, 2-way crossover study to assess pharmacodyamic and pharmacokinetic profiles following treatment with PL-ASA and EC-ASA administered under fasting condition at a single dose of 81 mg among the volunteers aged 50 to 75 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female non-smoking subjects between the ages of 18 to 75 years inclusive, without known medical conditions requiring treatment
* Consumes on average no more than 2 alcoholic drinks per day for 30 days prior to study

Exclusion Criteria:

* Abnormal baseline laboratory results
* Current prescribed use of aspirin, warfarin or other anticoagulants
* Use of other specific medications within 2 weeks of study start
* History of certain medical conditions
* Subject's platelets are unresponsive to arachidonic acid, as defined as <60% of aggregation as measured by light transmittance aggregometry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Acetylsalicylic acid and salicylic acid | 24 hours after dosing
  Presence of serum acetylsalicylic acid and salicylic acid

SECONDARY OUTCOMES:
Light transmittance aggregometry | 24 hours after dosing
  Effects on platelet function by light transmittance aggregometry

OTHER OUTCOMES:
Serum thromboxane B2 | 24 hours after dosing
  ncidence of aspirin responsiveness among study participants, measured by Inhibition of serum thromboxane B2 and thromboxane B2 levels
Adverse effects | 24 hours after dosing
  Safety, as indicated by any adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franchi, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida C, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Schneider DJ, Prats J, Fan W, Rollini F, Been L, Taatjes-Sommer HS, Bhatt DL, Deliargyris EN, Angiolillo DJ. Pharmacokinetic and pharmacodynamic profiles of a novel phospholipid-aspirin complex liquid formulation and low dose enteric-coated aspirin: results from a prospective, randomized, crossover study. J Thromb Thrombolysis. 2022 Oct;54(3):373-381. doi: 10.1007/s11239-022-02687-5. Epub 2022 Aug 29. PMID 36036856